CLINICAL TRIAL: NCT01041950
Title: Lumbar Drainage for Communicating Hydrocephalus After Intraventricular Hemorrhage: a Randomised, Controlled Trial(LUCAS-IVH: LUmbar CAtheter for Severe IntraVentricular Hemorrhage)
Brief Title: A Randomised Controlled Trial of Lumbar Drainage to Treat Communicating Hydrocephalus After Severe Intraventricular Hemorrhage
Acronym: LUCAS-IVH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University of Freiburg (Other)
Responsible Party: Principal Investigator, Dimitre Staykov, Priv.-Doz. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUCAS-IVH
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Intracerebral Hemorrhage; Obstructive Hydrocephalus
Keywords: intracerebral hemorrhage; intraventricular hemorrhage; hydrocephalus; Intracerebral hemorrhage with severe ventricular involvement and obstructive hydrocephalus
MeSH Terms: conditions — Cerebral Hemorrhage; Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar drainage (Experimental)
  Interventions: Procedure: Lumbar drainage
- Control (No Intervention)

INTERVENTIONS:
Procedure: Lumbar drainage — Lumbar CSF drainage is started after communication between the internal and external CSF-spaces is seen on CT.
  Arms: Lumbar drainage

SUMMARY:
The purpose of this study is to determine if usage of early lumbar drainage leads to less shunt surgery and less catheter associated complications in patients with communicating hydrocephalus after intracerebral hemorrhage with severe ventricular involvement.

DETAILED DESCRIPTION:
All patients requiring external ventricular drain (EVD) for treatment of acute obstructive hydrocephalus receive intraventricular fibrinolysis with rt-PA via the ventricular catheter. Lumbar drainage (LD) is inserted at a timepoint, when communication between the internal and the external CSF-spaces is recognizable on CT ("opening" of third and fourth ventricle and aqueduct).

ELIGIBILITY:
Inclusion Criteria:

* supratentorial intracerebral hemorrhage <60ml
* intraventricular hemorrhage with casting of the third and fourth ventricles
* obstructive hydrocephalus with need of external ventricular drainage
* GCS <9 on admission or within 48h of symptom onset
* admission within 48h of symptom onset
* preceding modified Rankin scale ≤3
* age 18-85 years

Exclusion Criteria:

* ICH related to oral anticoagulation, trauma, tumor, arteriovenous malformation, aneurysm, systemic thrombolysis or sinus thrombosis
* infratentorial hemorrhage
* pregnancy
* admission 48h after symptom onset
* preceding modified Rankin scale >3

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Requirement of permanent VP-shunt | 14 days
  if three attempts to clamp the EVD (control group) or LD (treatment group) fail, or overall extra-corporal drainage time exceeds 14 days, a VP-shunt is placed.

SECONDARY OUTCOMES:
Safety aspects | during hospital stay
  (i) catheter-associated infections (ii) fibrinolysis- and catheter-associated bleedings (iii)overdrainage and herniation
mortality and outcome | 3 and 6 months
  modified Rankin Scale 3 and 6 months after treatment, as well as in-hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Huttner, MD, Principal Investigator — Neurology Department, University of Erlangen-Nuremberg; Dimitre Staykov, MD, Principal Investigator — Neurology Department, University of Erlangen-Nuremberg; Jürgen Bardutzky, MD, Study Chair — University of Freiburg
Locations (1):
- Neurology Department, University of Erlangen-Nuremberg, Erlangen, Germany

REFERENCES:
- [Derived] Staykov D, Kuramatsu JB, Bardutzky J, Volbers B, Gerner ST, Kloska SP, Doerfler A, Schwab S, Huttner HB. Efficacy and safety of combined intraventricular fibrinolysis with lumbar drainage for prevention of permanent shunt dependency after intracerebral hemorrhage with severe ventricular involvement: A randomized trial and individual patient data meta-analysis. Ann Neurol. 2017 Jan;81(1):93-103. doi: 10.1002/ana.24834. PMID 27888608